CLINICAL TRIAL: NCT01658046
Title: Effects of Neuromuscular Electrical Stimulation as an Adjunct to Exercise Training in Stable COPD
Brief Title: Effects of Neuromuscular Electrical Stimulation as an Adjunct to Exercise Training in Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Deniz Inal-Ince, PhD, PT, Associated Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMES-COPD; Hacettepe University (Other: Hacettepe University)
Record Dates: First submitted 2012-07-31; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; exercise; neuromuscular electrical stimulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Endurance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMES group (Experimental): 10 weeks neuromuscular electrical stimulation plus endurance training and quadriceps strength training.
  Interventions: Other: Neuromuscular electrical stimulation; Other: Endurance training; Other: Quadriceps strength training
- Control group (Sham Comparator): 10 weeks sham neuromuscular electrical stimulation plus endurance training and quadriceps strength training.
  Interventions: Other: Endurance training; Other: Quadriceps strength training

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — Bilateral quadriceps NMES using a four-channel portable electrical stimulator. Biphasic symmetric constant current impulses with a pulse width 300 µs, a frequency of 50 Hz, and duty cycle of 10 s on and 20 s off was applied for 20 min per day, 2 days per week for 10 weeks.
  Arms: NMES group
Other: Endurance training — Endurance training consists of 30 minutes of aerobic exercise (15 minutes on treadmill and 15 minutes on stationary bicycle) at 80% of maximal heart rate
Other: Quadriceps strength training — Quadriceps resistance training was applied using free weights for 2 days per week for 10 weeks according to 1 repetition maximum, starting at 45% for two sets.

SUMMARY:
Skeletal muscle dysfunction impairs exercise capacity, quality of life and prognosis in chronic obstructive pulmonary disease (COPD). The purpose of this prospective randomized controlled study was to evaluate effects of Neuromuscular electrical stimulation (NMES) plus quadriceps muscle training (NMES group) and sham NMES plus quadriceps muscle training (control group) on muscle function, exercise capacity, health related quality of life, activities of daily living, and self-efficacy in patients with COPD who are eligible and able to participate in endurance training.

DETAILED DESCRIPTION:
Skeletal muscle dysfunction is common and impaires exercise capacity in patients with chronic obstructive pulmonary disease (COPD)Exercise training is the main component of the treatment of COPD.

Neuromuscular electrical stimulation (NMES) is successful in COPD patients who are unable to perform exercise training. The NMES has positive effect on peripheral muscle function, exercise capacity and breathlessness in activities of daily living in COPD patients who had an abnormal body composition or who were too dyspneic to leave their home. A nonrandomized uncontrolled study has shown that application of NMES at home for improved exercise capacity in patients with better-preserved muscle mass. Evidence from a preliminary study without applying sham NMES revealed that NMES applied as complementary to ambulatory respiratory rehabilitation program increased quadriceps strength, quality of life and six minute walk distance in severe to very severe patients.

Despite documented benefits of NMES in COPD patients, the place of NMES as an adjunct to pulmonary rehabilitation in COPD patients who were able to do regular endurance and strength training on is unknown. Therefore, the purpose of this study was to compare the effects of NMES plus quadriceps muscle training (NMES group) and sham NMES plus quadriceps muscle training (control group) on muscle function, dyspnea, fatigue, exercise capacity, health related quality of life, activities of daily living, and self-efficacy in patients with COPD who are eligible and able to participate in endurance training.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic obstructive pulmonary disease
* being 35-75 years of age
* being eligible to participate in endurance trainin
* no acute exacerbation in last month, no change in drugs and no usage of antibiotics in last three weeks

Exclusion Criteria:

* medical conditions which could place patient at risk during neuromuscular electrical stimulation and exercise training (orthophedic and neuromuscular disorders, metal implants in the lower limbs, advanced heart failure, aortic stenosis, deep venous thrombosis a cardiac pacemaker, >50 mmHg pulmonary artery pressure and/or an acute exacerbation of symtomps in the preceeding four weeks)
* being unable to understand the questionnaires and unable to cooparate.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Incremental shuttle walk test | 10 weeks
  The incremental shuttle walk test was performed in an enclosed corridor. Patients were required to walk back and forth, turning around two cones placed 9 meters apart making the shuttle distance 10 meters long. Patients followed the rhythm dictated by the audio signal.

SECONDARY OUTCOMES:
Endurance shuttle walk test | 10 weeks
  An endurance shuttle walk test was used to measure endurance walking capacity. The endurance shuttle walk test was performed 85% of peak oxygen consumption as predicted from the incremental shuttle walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, PhD, PT, Principal Investigator — Hacettepe University
Locations (1):
- Ataturk Chest Diseases and Thoracic Surgery Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Tasdemir F, Inal-Ince D, Ergun P, Kaymaz D, Demir N, Demirci E, Egesel N. Neuromuscular electrical stimulation as an adjunct to endurance and resistance training during pulmonary rehabilitation in stable chronic obstructive pulmonary disease. Expert Rev Respir Med. 2015 Aug;9(4):493-502. doi: 10.1586/17476348.2015.1068691. Epub 2015 Jul 15. PMID 26175226